CLINICAL TRIAL: NCT00827918
Title: A Phase IIa, Randomized, Multicenter, Double-Blind, Active Comparator- and Placebo-Controlled, Clinical Trial to Study the Safety and Efficacy of MK8998 in Acutely Psychotic Patients With Schizophrenia
Brief Title: A Study to Test the Safety and Efficacy of MK-8998 in Acutely Psychotic Participants With Schizophrenia (MK-8998-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8998-004; 2009_519
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia
Keywords: Acute Exacerbation of Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MK-8998 (Experimental): MK-8998, 6 mg twice a day (BID) for Days 1 to 7, and 8 mg BID thereafter for a 4-week total treatment period
  Interventions: Drug: MK-8998
- Olanzapine (Active Comparator): Olanzapine, 5 mg BID for Day 1 to 7, and 15 mg (5 mg in the morning and 10 mg in the evening) thereafter for a 4-week total treatment period
  Interventions: Drug: Comparator: Olanzapine
- Placebo (Placebo Comparator): Placebo Comparator to MK-8998 or olanzapine
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK-8998 — MK-8998 6 mg capsules twice daily with food on Days 1 through 7. On Day 8, dosage will be increased to 8 mg capsules twice daily. Treatment period is 4 weeks. There will be a period of time when all participants will receive placebo.
  Arms: MK-8998
Drug: Comparator: Olanzapine — Olanzapine 5 mg tablets twice daily with food on Days 1 through 7. On Day 8, dosage will be increased to 5 mg tablets in the morning and 10 mg tablets in the evening. Treatment period is 4 weeks. There will be a period of time when all participants will receive placebo.
  Arms: Olanzapine
Drug: Comparator: Placebo — Placebo tablets matching olanzapine tablets and MK-8998 capsules
  Arms: Placebo

SUMMARY:
A study to evaluate the safety and efficacy of treatment with MK-8998 as compared to placebo and olanzapine for acutely psychotic patients with schizophrenia. The primary hypothesis is that in participants undergoing an acute psychotic episode of schizophrenia, MK-8998 6 to 8 mg twice daily is superior to placebo in the treatment of symptoms of schizophrenia as measured by the mean change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score at Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age is 18 to 55
* Patient meets DSM-IV/DSM-IV-TR criteria for a primary diagnosis of schizophrenia
* The duration of the patients schizophrenia diagnosis must be greater than 1 year
* Patient has an acute exacerbation of psychotic symptoms (of at least 3 days but no longer than 6 weeks) and marked deterioration of function

Exclusion Criteria:

* Patient currently has a clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorder that would pose a risk to the patient in the opinion of the investigator if they were to participate in the study or that might confound the results of the study
* The patient has evidence of acute hepatitis, clinically significant chronic hepatitis, or impaired hepatic function
* The patient has a chronic organic disease of the central nervous system (other than schizophrenia) such as, tumors, inflammation, active seizure disorder, vascular disorder, Parkinson's disease, Alzheimer's disease or other forms of dementia, myasthenia gravis, or other degenerative processes. In addition, patients must not have a history of mental retardation or persistent neurological symptoms attributable to serious head injury
* Patient has a history of alcohol/drug dependence within 3 months or alcohol/drug abuse within 1 month of screening. Exceptions include caffeine and nicotine abuse/dependence
* Patient has a history of hypersensitivity to olanzapine OR poor response to olanzapine in the last 2 years OR intolerable side effects due to olanzapine OR patients current psychotic relapse occurred while consistently taking a therapeutic dose (10 mg or more) of olanzapine OR olanzapine is medically contradicted
* Patient is refractory to antipsychotic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Egan MF, Zhao X, Smith A, Troyer MD, Uebele VN, Pidkorytov V, Cox K, Murphy M, Snavely D, Lines C, Michelson D. Randomized controlled study of the T-type calcium channel antagonist MK-8998 for the treatment of acute psychosis in patients with schizophrenia. Hum Psychopharmacol. 2013 Mar;28(2):124-33. doi: 10.1002/hup.2289. PMID 23532746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female inpatients who were experiencing an acute exacerbation of schizophrenia were randomized at 21 sites worldwide.
Pre-assignment Details: Participants who met entry criteria were washed out of psychotropic medication and then entered a single-blind, in-patient, 3-day to 7-day, placebo lead-in period.
Groups:
- MK-8998: MK-8998, 6 mg twice a day (BID) on Days 1 to 7, and 8 mg BID thereafter for a 4-week total treatment period
- Olanzapine: Olanzapine, 5 mg BID on Day 1 to 7, and 15 mg (5 mg in the morning and 10 mg in the evening) thereafter for a 4-week total treatment period
- Placebo Comparator: Placebo Comparator to MK-8998 or olanzapine
Period: Overall Study
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Started | 86 | 47 | 83
Completed | 58 | 38 | 62
Not Completed | 28 | 9 | 21
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Lack of Efficacy | 16 | 4 | 15
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Progressive Disease | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator | Total
Number analyzed (Participants) | 86 | 47 | 83 | 216
Age, Continuous [Mean (Full Range); unit: years] | 37.4 [21 to 55] | 36.1 [20 to 55] | 36.4 [22 to 54] | 36.8 [20 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 23 | 30 | 90
  Male | 49 | 24 | 53 | 126

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) at Week 4
Description: PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. PANSS measure is composed of 3 scales: Positive scale, Negative scale, and General Psychopathology scale. Positive scale assesses hallucinations, delusions and related symptoms; Negative scale assesses emotional withdrawal, lack of motivation, and similar symptoms; and General Psychopathology scale addresses other symptoms such as anxiety, somatic concern and disorientation. The PANSS has 30 items in its 3 scales and an anchored Likert scale from 1 to 7 is used to score each item. Values of 2 and above indicate the presence of progressively more severe symptoms. The Positive scale has 7 items with a score from 7 to 49, the Negative scale has 7 items with a score from 7 to 49, and the General Psychopathology scale has 16 items with a score from 16 to 112. A total score is the sum of the 3 scores for the 3 scales.
Time Frame: Baseline and Week 4
Population: Randomized participants with any PANSS measurements between Baseline and Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 81 | 45 | 78
Units on a scale | -13.3 [-17.9 to -8.7] | -17.0 [-22.8 to -11.1] | -12.7 [-17.2 to -8.2]
Statistical Analysis 1: Comparison: MK-8998 vs Placebo Comparator; Test type: Superiority or Other; p = 0.8590, Difference in the Least Squares Mean; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-7.0 to 5.8]
Statistical Analysis 2: Comparison: Olanzapine vs Placebo Comparator; Test type: Superiority or Other; p = 0.2534, Difference in the Least Squares Mean; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-11.7 to 3.1]

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the study drug.
Time Frame: Up to 6 Weeks
Population: All participants included in the All Patients as Treated (APaT) population received at least one dose of study treatment and were evaluated for safety.
Measure: Number; unit: Participants
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 86 | 47 | 83
Participants | 41 | 23 | 33

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the study drug.
Time Frame: Up to 4 Weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 86 | 47 | 83
Participants | 9 | 1 | 1

4. Secondary Outcome: Percentage of Participants With Response at Week 4
Description: Responders were defined as participants who demonstrated ≥ 20% improvement from baseline on the PANSS total score. PANSS measure is composed of 3 scales: Positive scale, Negative scale, and General Psychopathology scale. Positive scale assesses hallucinations, delusions and related symptoms; Negative scale assesses emotional withdrawal, lack of motivation, and similar symptoms; and General Psychopathology scale addresses other symptoms such as anxiety, somatic concern and disorientation. The PANSS has 30 items in its 3 scales and an anchored Likert scale from 1 to 7 is used to score each item. Values of 2 and above indicate the presence of progressively more severe symptoms. The Positive scale has 7 items with a score from 7 to 49, the Negative scale has 7 items with a score from 7 to 49, and the General Psychopathology scale has 16 items with a score from 16 to 112. A total score is the sum of the 3 scores for the 3 scales.
Time Frame: Week 4
Population: Randomized participants with a PANSS measurement at Week 4.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 54 | 36 | 58
Percentage of participants | 57.4 | 66.7 | 48.3
Statistical Analysis 1: Comparison: MK-8998 vs Placebo Comparator; Test type: Superiority or Other; p = 0.4976, Generalized linear mixed analysis model; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.62 to 2.64]
Statistical Analysis 2: Comparison: Olanzapine vs Placebo Comparator; Test type: Superiority or Other; p = 0.0653, Generalized linear mixed analysis model; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.95 to 5.09]

5. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Severity of Illness Scale (CGI-S) at Week 4
Description: CGI-S is a commonly used measure of symptom severity in treatment studies of participants with mental disorders. CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill.
Time Frame: Baseline and Week 4
Population: Randomized participants with any CGI-S measurements between baseline and Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 81 | 45 | 78
Units on a scale | -0.9 [-1.2 to -0.7] | -0.8 [-1.2 to -0.5] | -0.9 [-1.1 to -0.6]
Statistical Analysis 1: Comparison: MK-8998 vs Placebo Comparator; Test type: Superiority or Other; p = 0.8199, Constrained longitudinal data analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 2: Comparison: Olanzapine vs Placebo Comparator; Test type: Superiority or Other; p = 0.9486, Constrained longitudinal data analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]

6. Secondary Outcome: Mean Change From Baseline in PANSS Positive Subscale at Week 4
Description: PANSS Positive scale assesses hallucinations, delusions and related symptoms. The Positive scale has 7 items with an anchored Likert scale from 1 to 7 to score each item. Values of 2 and above indicate the presence of progressively more severe symptoms. A total score ranges from 7 to 49.
Time Frame: Baseline and Week 4
Population: Randomized participants with any PANSS positive subscale measurements between baseline and Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 81 | 45 | 78
Units on a scale | -4.2 [-5.6 to -2.8] | -5.6 [-7.4 to -3.8] | -4.2 [-5.6 to -2.9]
Statistical Analysis 1: Comparison: MK-8998 vs Placebo Comparator; Test type: Superiority or Other; p = 0.9937, Constrained longitudinal data analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-2.0 to 2.0]
Statistical Analysis 2: Comparison: Olanzapine vs Placebo Comparator; Test type: Superiority or Other; p = 0.2406, Constrained longitudinal data analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.6 to 0.9]

7. Secondary Outcome: Mean Change From Baseline in PANSS Negative Subscale at Week 4
Description: PANSS Negative scale assesses emotional withdrawal, lack of motivation, and similar symptoms. The Negative scale has 7 items with an anchored Likert scale from 1 to 7 to score each item. Values of 2 and above indicate the presence of progressively more severe symptoms. A total score ranges from 7 to 49.
Time Frame: Baseline and Week 4
Population: Randomized participants with any PANSS negative subscale measurements between baseline and Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Number analyzed (Participants) | 81 | 45 | 78
Units on a scale | -3.3 [-4.5 to -2.2] | -3.1 [-4.5 to -1.6] | -2.9 [-4.0 to -1.8]
Statistical Analysis 1: Comparison: MK-8998 vs Placebo Comparator; Test type: Superiority or Other; p = 0.5953, Constrained longitudinal data analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.0 to 1.2]
Statistical Analysis 2: Comparison: Olanzapine vs Placebo Comparator; Test type: Superiority or Other; p = 0.8567, Constrained longitudinal data analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.0 to 1.6]

ADVERSE EVENTS:
Time Frame: Up to 6 Weeks
Arm/Group | MK-8998 | Olanzapine | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/47 | 1/83
Other Adverse Events (participants affected / at risk) | 19/86 | 14/47 | 11/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8998 (N=86) | Olanzapine (N=47) | Placebo Comparator (N=83)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8998 (N=86) | Olanzapine (N=47) | Placebo Comparator (N=83)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 3 (4)
Somnolence (Nervous system disorders) | 2 (2) | 3 (8) | 1 (1)
Insomnia (Psychiatric disorders) | 13 (14) | 5 (6) | 7 (8)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.